CLINICAL TRIAL: NCT05630911
Title: The Effects of Conscious Movement Processing on Postural Stability and Muscle Efficiency While Standing in a Challenging Environment by Older Adults at Risk of Falling in Hong Kong: Implications for Rehabilitation.
Brief Title: Conscious Movement Processing, Postural Stability and Muscle Efficiency in Older Adults
Status: Recruiting | Type: Observational
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Other Study IDs: 15600322
Record Dates: First submitted 2022-11-18; First posted 2022-11-30 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Fall Injury; Postural; Defect; Old Age; Debility
Keywords: Older Adults in Hong Kong; Conscious Movement Processing; Postural Stability; Muscle Efficiency; Attentional Focus
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High Reinvestor Group (HRG): Participants will be invited to complete a series of standing balance trials. The trials will involve participants standing in three different positions on a foam surface (i.e., Airex balance pad elite with a dimension of 16.1" width x 19.7" length x 2.4" height, or equivalent).The three different standing positions will be: wide-base standing on foam (WBF), narrow-base standing on foam (NBF), and tandem standing on foam (TAF) (i.e., low-level of task difficulty, moderate-level of task difficulty, and high-level of task difficulty, respectively). For each standing position, participants will be required to perform two consecutive standing balance trials, with a 1-minute rest break in between.
  Interventions: Other: Standing tasks with different task difficulty
- Low Reinvestor Group (LRG): Participants will be invited to complete a series of standing balance trials. The trials will involve participants standing in three different positions on a foam surface (i.e., Airex balance pad elite with a dimension of 16.1" width x 19.7" length x 2.4" height, or equivalent).The three different standing positions will be: wide-base standing on foam (WBF), narrow-base standing on foam (NBF), and tandem standing on foam (TAF) (i.e., low-level of task difficulty, moderate-level of task difficulty, and high-level of task difficulty, respectively). For each standing position, participants will be required to perform two consecutive standing balance trials, with a 1-minute rest break in between.
  Interventions: Other: Standing tasks with different task difficulty

INTERVENTIONS:
Other: Standing tasks with different task difficulty — The three different standing positions will include wide-base standing on foam (WBF) with low-level of task difficulty, narrow-base standing on foam (NBF) with moderate-level of task difficulty, and tandem standing on foam (TAF) with high-level of task difficulty.

SUMMARY:
This study aims to address critical knowledge gaps by investigating the effects of trait conscious movement processing propensity on real-time (state) conscious movement processing propensity, postural stability, and muscle efficiency in older adults at risk of falling in Hong Kong with high and low trait conscious movement processing propensities, while standing in a challenging environment with different levels of standing task difficulties. The study results would contribute to our scientific understanding of the mechanisms of conscious movement processing in older adults while maintaining standing balance in a challenging environment. It could inform the follow-up investigations for the development of the most appropriate psychomotor standing balance re-education intervention in rehabilitation so as to mitigate the effect of conscious movement processing and the risk of falling in older adults. The findings from the proposed research could ultimately help improve the outcome of fall rehabilitation programmes and reduce the impact of falls in the older adults in Hong Kong.

ELIGIBILITY:
Inclusion Criteria:

* 65 years old or above;
* able to stand independently without a walking aid.

Exclusion Criteria:

* a history of any major cerebrovascular and/or neurological disorders (e.g., stroke, Parkinson's disease);
* a history of a major fall event within the past year;
* the existence of an unstable medical or mobility condition that could affect safety in this study;
* a score of 23/30 or below in the Chinese version of Mini-Mental State Examination (MMSE-C);
* a static visual acuity poorer than 20/40 vision (examined by the Tumbling-E eye chart).

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: The recruitment of older adult participants (N = 132) will take place at collaborating rehabilitative and elderly community centres in Hong Kong through convenience sampling. Potential participants will be screened for eligibility according to the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Real-time (state) conscious movement processing propensity | Day 0
  It will be measured by the Alpha2 electrocephalogram (EEG) T3-Fz coherence.

SECONDARY OUTCOMES:
Postural stability | Day 0
  It will be measured by the 3-D motion capture system to identify the postural sway in the unit of millimeter (mm) or the postural sway velocity in the unit of meter per second (m/s).
Muscle efficiency | Day 0
  It will be measured by the surface electromyography (EMG).
Functional mobility | Day 0
  It will be measured by the Timed 'Up & Go' (TUG) test.
Balance ability | Day 0
  It will be measured by the Berg Balance Scale. The minimum value of the scale is 0 and the maximum value is 56. Higher score represents better balance ability.
Fear of falling | Day 0
  It will be measured by the Falls Efficacy Scale International. The minimum value of the scale is 16 and the maximum value is 64. Higher score represents higher fear of falling.
Trait conscious movement processing propensity | Day 0
  It will be measured by the the Chinese version of the Movement-Specific Reinvestment Scale. The minimum value of the scale is 10 and the maximum value is 60. Higher score represents higher trait conscious movement processing propensity.
Perceived standing task difficulty | Day 0
  It will be measured by the Visual Analog Scale. The minimum value of the scale is 0 and the maximum value is 100. Higher score represents higher perceived standing task difficulty.

CONTACTS AND LOCATIONS:
Overall Officials: Thomson Wong, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No